CLINICAL TRIAL: NCT06287294
Title: An Investigation Into Taste Problems Associated With Xerostomia in Patients With Advanced Cancer
Status: Recruiting | Type: Observational
Sponsor: Our Lady's Hospice and Care Services (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, Our Lady's Hospice and Care Services
Other Study IDs: RS23-042
Record Dates: First submitted 2023-11-20; First posted 2024-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Taste, Altered; Xerostomia; Neoplasms
MeSH Terms: conditions — Dysgeusia; Xerostomia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taste problems and xerostomia (dry mouth) are common among patients with advanced cancer. These symptoms can affect the pleasure of eating and drinking, reduce dietary intake, cause low mood, and a lower quality of life. This study will explore the relationship between dry mouth and taste problems in patients with advanced cancer.

DETAILED DESCRIPTION:
Patients with advanced cancer often develop taste disturbances. A recent literature review reported a median prevalence of 55%, with prevalence ranging from 27-93%. Studies have shown taste disturbance is usually a persistent symptom, is often 'moderate-to-severe' in intensity, and is often associated with significant distress. Taste disturbance may have a major impact on the experience and pleasure associated with eating and drinking. Taste disturbance may have a major impact on nutritional intake. It may be associated with low mood / depression, social isolation, and an impaired quality of life.

There is limited data available on the aetiology of taste disturbances in patients with advanced cancer, although one group of researchers reported an association between the severity of xerostomia (subjective sensation of dry mouth) and the severity of taste disturbance. Several studies have identified xerostomia and taste disturbance in symptom clusters.

Xerostomia (dry mouth) is defined as the subjective complaint of dry mouth. The prevalence of xerostomia in patients with advanced cancer has been reported to be >80%. It is the most common oral symptom in patients with advanced cancer. Xerostomia is often a distressing symptom, and is associated with a number of complications including oral discomfort, lip discomfort, cracking of lips, taste disturbances, difficulty chewing, difficulty swallowing, decreased intake of nutrition, oesophagitis, difficulty speaking, poor oral hygiene, halitosis, dental caries, salivary gland infections, oral candidiasis, pneumonia, dental demineralisation (causing dental sensitivity), denture fitting problems, oesophagitis, sleep disturbance, embarrassment, anxiety, depression, and social isolation.

The aforementioned literature review identified the need for observational studies to determine the prevalence, clinical features, "risk factors" and aetiologies for taste disturbance- this data would facilitate targeted screening for the problem. Studies have shown that taste disturbances and xerostomia often co-exist. To the researcher's knowledge, there no evidence on the effect of xerostomia or its treatment on taste problems. This study will explore the relationship between xerostomia and taste problems in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnosis of locally advanced or metastatic cancer
* Referred to palliative care/oncology services
* Dry mouth rated 'moderate' or worse over previous 2-week period
* Taste problems rated 'moderate' or worse over previous 2-week period
* Good understanding of English

Exclusion Criteria:

* Cognitive impairment (unable to provide consent / complete questionnaire)
* Dry mouth precedes cancer diagnosis.
* Taste problems precedes cancer diagnosis.
* Head and neck surgery
* Head and neck radiotherapy
* Salivary gland disorders (e.g., Sjogren's Syndrome)
* In the 'Deteriorating' or 'Terminal' Phase of illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently under the care of oncology or palliative care who have an incurable cancer. Patients will be identified by the clinical teams at the study sites, informed about the study, and (if interested in taking part in the study) referred to the research team.
  Participants will be screened for inclusion by asking, "1. Over the last 2 weeks have you experienced having a dry mouth? 2. Over the past 2 weeks have you experienced taste problems?" If yes to either question, "How severe was it? (Options- Slight/Moderate/Severe/Very severe)". Patients must score as moderate/severe/very severe.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure the prevalence of taste problems in patients with advanced cancer with a dry mouth using the Oral Symptom Assessment Scale (questionnaire) | December 2025
  To measure the prevalence of taste problems in patients with advanced cancer who have a dry mouth using the validated Oral Symptom Assessment Scale, which is a 20 question questionnaire which asks about the presence of symptoms in the previous week, the frequency of the symptoms, the severity of the symptoms, and the amount of distress/"bothersomeness" caused by the symptoms.
To identify an association of any other oral symptoms present in patients with taste problems and dry mouth who have advanced cancer using the Oral Symptom Assessment Scale (questionnaire) | December 2025
  To identify an association of any other oral symptoms present in patients with taste problems and dry mouth who have advanced cancer using the Oral Symptom Assessment Scale (questionnaire) which asks about the presence of symptoms in the previous week, the frequency of the symptoms, the severity of the symptoms, and the amount of distress/"bothersomeness" caused by the symptoms.
To characterise the taste disturbances i.e. to identify reduced taste, heightened taste, altered taste or no taste using the Taste Questionnaire in Palliative Care (questionnaire) and Waterless Empirical Taste Test (objective taste test) | December 2025
  To characterise the taste disturbances i.e. for reduced taste, heightened taste, altered taste or no taste using the Taste Questionnaire in Palliative Care, which is a 16 question questionnaire which asks about the presence of taste problems in the previous fortnight, the frequency of the symptoms, the severity of the symptoms, and the amount of distress/"bothersomeness" caused by these symptoms. An objective taste test, the Waterless Empirical Taste Test will also be used. This is comprised of taste strips with monomer cellulose pads impregnated with solutions dried of sucrose, citric acid, sodium chloride, caffeine, monosodium glutamate, or no stimulus. The participant is instructed to move the cellulose pad of each strip around the mouth for 5-10 seconds, and to identify the taste quality or to indicate that no taste can be perceived.
To identify what impact taste problems are having on patients dietary intake using the Taste Questionnaire in Palliative Care (questionnaire). | December 2025
  To identify the impact taste problems are having on patients dietary intake using the Taste Questionnaire in Palliative Care (questionnaire) which is a 16 question questionnaire which asks about the presence of taste problems and xerostomia in the previous fortnight, the frequency of the symptoms, the severity of the symptoms, and the amount of distress/"bothersomeness" caused by these symptoms.
To identify what impact taste problems are having on patients quality of life using the Taste Questionnaire in Palliative Care (questionnaire). | December 2025
  To identify the impact taste problems are having on patients quality of life using the Taste Questionnaire in Palliative Care (questionnaire) which is a 16 question questionnaire which asks about the presence of taste problems and xerostomia in the previous fortnight, the frequency of the symptoms, the severity of the symptoms, and the amount of distress/"bothersomeness" caused by these symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, FRCP, Principal Investigator — Our Lady's Hospice and Care Services
Locations (1):
- Our Lady's Hospice and Care Services, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Hannon M, Shaw A, Connolly M, Davies A. Taste disturbance in patients with advanced cancer: a scoping review of clinical features and complications. Support Care Cancer. 2023 Sep 6;31(10):562. doi: 10.1007/s00520-023-08012-x. PMID 37672147
- [Background] Davies A, Buchanan A, Todd J, Gregory A, Batsari KM. Oral symptoms in patients with advanced cancer: an observational study using a novel oral symptom assessment scale. Support Care Cancer. 2021 Aug;29(8):4357-4364. doi: 10.1007/s00520-020-05903-1. Epub 2021 Jan 8. PMID 33416995
- [Background] McGettigan N, Dhuibhir PU, Barrett M, Sui J, Balding L, Higgins S, O'Leary N, Kennedy A, Walsh D. Subjective and Objective Assessment of Taste and Smell Sensation in Advanced Cancer. Am J Hosp Palliat Care. 2019 Aug;36(8):688-696. doi: 10.1177/1049909119832836. Epub 2019 Mar 3. PMID 30827119
- [Background] Twycross RG, Lack SA (1986) Control of alimentary symptoms in far advanced cancer. Churchill Livingstone, Edinburgh
- [Background] Kirkova J, Walsh D, Rybicki L, Davis MP, Aktas A, Tao Jin, Homsi J. Symptom severity and distress in advanced cancer. Palliat Med. 2010 Apr;24(3):330-9. doi: 10.1177/0269216309356380. Epub 2009 Dec 16. PMID 20015920
- [Background] Webber K, Davies AN, Leach C, Waghorn M. Symptom prevalence and severity in palliative cancer medicine. BMJ Support Palliat Care. 2023 Dec 7;13(e2):e270-e272. doi: 10.1136/bmjspcare-2020-002357. PMID 34130997
- [Background] Hutton JL, Baracos VE, Wismer WV. Chemosensory dysfunction is a primary factor in the evolution of declining nutritional status and quality of life in patients with advanced cancer. J Pain Symptom Manage. 2007 Feb;33(2):156-65. doi: 10.1016/j.jpainsymman.2006.07.017. PMID 17280921
- [Background] Rydholm M, Strang P. Physical and psychosocial impact of xerostomia in palliative cancer care: a qualitative interview study. Int J Palliat Nurs. 2002 Jul;8(7):318-23. doi: 10.12968/ijpn.2002.8.7.10671. PMID 12165715
- [Background] Davies AN, Broadley K, Beighton D. Xerostomia in patients with advanced cancer. J Pain Symptom Manage. 2001 Oct;22(4):820-5. doi: 10.1016/s0885-3924(01)00318-9. PMID 11576798
- [Background] Tsai JS, Wu CH, Chiu TY, Chen CY. Significance of symptom clustering in palliative care of advanced cancer patients. J Pain Symptom Manage. 2010 Apr;39(4):655-62. doi: 10.1016/j.jpainsymman.2009.09.005. Epub 2010 Mar 11. PMID 20226623
- [Background] Walsh D, Rybicki L. Symptom clustering in advanced cancer. Support Care Cancer. 2006 Aug;14(8):831-6. doi: 10.1007/s00520-005-0899-z. Epub 2006 Feb 16. PMID 16482450
- [Background] Hopcraft MS, Tan C. Xerostomia: an update for clinicians. Aust Dent J. 2010 Sep;55(3):238-44; quiz 353. doi: 10.1111/j.1834-7819.2010.01229.x. PMID 20887509